CLINICAL TRIAL: NCT03605641
Title: An Open-Label, Single-Center Clinical Trial to Evaluate Selected Constituents in the Exhaled Breath and Room Air From the Use of E-vapor Products and Conventional Cigarettes Studied Under Residential, Office and Hospitality Environmental Conditions
Brief Title: Study to Evaluate Constituents in Exhaled Breath and Room Air From Use of E-vapor Products and Conventional Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juul Labs, Inc. (Industry)
Collaborators: Inflamax Research Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 755-00045
Record Dates: First submitted 2018-07-16; First posted 2018-07-30 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2018-12

CONDITIONS: Second Hand Tobacco Smoke
Keywords: E-Cigarettes; Conventional Cigarettes; JUUL; VUSE
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- JUUL electronic cigarette (Experimental): JUUL electronic cigarette. Virginia Tobacco 5% tobacco-derived nicotine.
  Interventions: Other: JUUL
- VUSE Solo electronic cigarette (Active Comparator): Reynolds American International VUSE Solo electronic cigarette. Original flavor 4.8% tobacco-derived nicotine.
  Interventions: Other: VUSE Solo
- Conventional cigarette (Active Comparator): Canadian purchased, store bought (not hand-rolled) conventional full-flavored cigarettes of subjects' preference.
  Interventions: Other: Conventional Cigarette

INTERVENTIONS:
Other: JUUL — JUUL Virginia Tobacco
  Arms: JUUL electronic cigarette
Other: VUSE Solo — VUSE SOLO Original
  Arms: VUSE Solo electronic cigarette
Other: Conventional Cigarette — Subject preferred conventional cigarette
  Arms: Conventional cigarette

SUMMARY:
An open-label, single center, three-arm observational study to examine emissions from e-cigarettes versus conventional cigarettes under three environmental settings of typical residential, office and hospitality facilities.

DETAILED DESCRIPTION:
Specific constituents will be measured in exhaled breath samples (EBS) from adult e-vapor product users and smokers when they are using e-vapor products or smoking conventional cigarettes. These constituents and particle counts (PC), will be measured in the room air samples (RAS) collected in the environmental exposure chamber (EEC) where adult e-cigarette users and smokers are using electronic cigarettes or smoking conventional cigarettes.

All subjects will undergo a Screening Visit to assess if they meet study eligibility criteria. If all eligibility criteria are met and the subject signs informed consent, the subject will be assigned to one of three groups: Group I (JUUL), Group II (VUSE Solo), or Group III (Conventional Cigarettes).

All three Groups will be sequentially observed in environmental settings 1 (residential), 2 (office), and 3 (hospitality). The observation period allocated for each environmental setting will be 2-days and 2-overnights for Groups I and II, and 1-day and 1-overnight for Group III. Each observation period will be referred to as a "Clinic Visit".

Subjects will move on to subsequent Environment Settings (Clinic Visits 2 or 3) after completion of the previous Clinic Visit (1 or 2).

Subjects must return to the clinic for Clinic Visit 1 within 60 days of the Screening Visit. Clinic Visit 2 must occur 7 ± 2 days after the Clinic Visit 1, and Clinic Visit 3 must occur 7 ± 2 days after Clinic Visit 2.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria before being enrolled into the study. Subjects must:

1. Be informed of the nature of the study and agree to and are able to read, review, and sign the informed consent document (in English) prior to the first study procedure. The Investigator must be satisfied that the volunteer has the ability to read and communicate in English in order to participate in the study.
2. Subjects screened as a part of an IRB-approved General Screening Protocol at the CRO site may be included in this study without additional Screening procedures provided all the required Screening procedures have been performed within 60 days prior to Clinic Visit 1.
3. Be a healthy male or female volunteer aged 21 - 65 years at the time of Screening Visit.
4. Have a positive urine cotinine result at Screening (Screening Visit) of >200 ng/ml.
5. Be judged by the Investigator to be in good general health as documented by the medical history, physical examination (including but may not be limited to an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems), vital sign assessments, 12-lead electrocardiogram (ECG), clinical laboratory assessments, and by general observations. Any abnormalities or deviations outside the normal ranges for any clinical testing (laboratory tests, ECG, vital signs) can be repeated at the discretion of the Investigator and judged to be not clinically significant for study participation.
6. Agree to abide by the study restrictions and return for the required assessments.
7. Have a self-reported daily conventional cigarette consumption rate of a minimum of 10 cigarettes per day for a minimum of 3 months prior to Screening Visit.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria will not be enrolled in the study.

Subjects must not:

1. Report receiving any investigational product within 30 days prior to Screening (Screening Visit).
2. Report any presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, urologic, gastrointestinal, hepatic, immunologic, hematologic, endocrine, oncologic or neurologic system(s) or psychiatric disease as determined by the Investigator.
3. Have any clinically significant results from laboratory tests, physical examinations, vital signs assessments, and electrocardiograms, as judged by the Investigator.
4. Report a clinically significant illness during the 30 days prior to enrollment, as determined by the Investigator.
5. Report a history of drug or alcohol addiction or abuse within the past 1 year.
6. Have positive screen for alcohol or drugs of abuse at Screening (Screening Visit) or check-in at Clinical Visit 1.
7. Have positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (anti-HCV).
8. Have body mass index (BMI) greater than 40 kg/m2 or less than 18 kg/m2 at Screening (Screening Visit).
9. Have used prescription anti-diabetic medication and/or insulin therapy within 12 months of Screening (Screening Visit).
10. Have taken medication for depression or asthma within 6 months of Screening (Screening Visit).
11. Have used prescription or over-the-counter bronchodilator medication (eg, inhaled or oral β-agonists) within 6 months of Screening (Screening Visit).
12. Be breast-feeding or pregnant female subjects (confirmed by a positive pregnancy test). Female subjects, who are considered women of child bearing potential (WOCBP) and sexually active, must be willing and able to use an acceptable method of contraception from Screening (Screening Visit) through the end of the study.
13. Be allergic to propylene glycol or glycerin.
14. Be or have a first-degree relative (ie, parent, sibling or child) be a current employee of the Sponsor or Site.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2018-12-02 (Actual)

PRIMARY OUTCOMES:
Exhaled Breath Sample (EBS) - Nicotine | Clinic Visit (JUUL/VUSE: 2 days and 2 overnights; conventional cigarette: 1 day and 1 overnight)
  Absolute change from baseline in nicotine levels in the EBS of subjects who use JUUL, VUSE Solo, or conventional cigarettes.
Exhaled Breath Sample (EBS) - Propylene glycol | Clinic Visit (JUUL/VUSE: 2 days and 2 overnights; conventional cigarette: 1 day and 1 overnight)
  Absolute change from baseline in propylene glycol levels in the EBS of subjects who use JUUL, VUSE Solo, or conventional cigarettes.
Exhaled Breath Sample (EBS) - Vegetable Glycerin | Clinic Visit (JUUL/VUSE: 2 days and 2 overnights; conventional cigarette: 1 day and 1 overnight)
  Absolute change from baseline in vegetable glycerin levels in the EBS of subjects who use JUUL, VUSE Solo, or conventional cigarettes.
Exhaled Breath Sample (EBS) - Carbonyls | Clinic Visit (JUUL/VUSE: 2 days and 2 overnights; conventional cigarette: 1 day and 1 overnight)
  Absolute change from baseline in carbonyl levels in the EBS of subjects who use JUUL, VUSE Solo, or conventional cigarettes. Carbonyl compounds include: formaldehyde, acetaldehyde, and acrolein.
Room Air Sample (RAS) - Nicotine | Clinic Visit (JUUL/VUSE: 2 days and 2 overnights; conventional cigarette: 1 day and 1 overnight)
  Absolute change from baseline in nicotine levels in the room air when subjects use JUUL or VUSE Solo over 4-hour prescribed conditions and JUUL, VUSE Solo, or conventional cigarettes over 4-hour ad libitum conditions.
Room Air Sample (RAS) - Propylene glycol | Clinic Visit (JUUL/VUSE: 2 days and 2 overnights; conventional cigarette: 1 day and 1 overnight)
  Absolute change from baseline in propylene glycol levels in the room air when subjects use JUUL or VUSE Solo over 4-hour prescribed conditions and JUUL, VUSE Solo, or conventional cigarettes over 4-hour ad libitum conditions.
Room Air Sample (RAS) - Vegetable Glycerin | Clinic Visit (JUUL/VUSE: 2 days and 2 overnights; conventional cigarette: 1 day and 1 overnight)
  Absolute change from baseline in vegetable glycerin levels in the room air when subjects use JUUL or VUSE Solo over 4-hour prescribed conditions and JUUL, VUSE Solo, or conventional cigarettes over 4-hour ad libitum conditions.
Room Air Sample (RAS) - Carbonyls | Clinic Visit (JUUL/VUSE: 2 days and 2 overnights; conventional cigarette: 1 day and 1 overnight)
  Absolute change from baseline in carbonyl levels in the room air when subjects use JUUL or VUSE Solo over 4-hour prescribed conditions and JUUL, VUSE Solo, or conventional cigarettes over 4-hour ad libitum conditions. Carbonyl compounds include: formaldehyde, crotonaldehyde, o-tolualdehyde, acetaldehyde, butyraldehyde (butanal), m&p-tolualdehyde, acetone, benzaldehyde, propionaldehyde, isovaleraldehyde, hexanaldehyde (aka hexaldehyde), valeraldehyde, 2, 5-dimethylbenzaldehyde, methyl ethyl ketone (MEK), acrolein.
Room Air Sample (RAS) - Volatile organic compounds | Clinic Visit (JUUL/VUSE: 2 days and 2 overnights; conventional cigarette: 1 day and 1 overnight)
  Absolute change from baseline in volatile organic compound levels in the room air when subjects use JUUL or VUSE Solo over 4-hour prescribed conditions and JUUL, VUSE Solo, or conventional cigarettes over 4-hour ad libitum conditions. Volatile organic compounds include: 1,3-butadiene, Benzene, isoprene, toluene, furan, ethylene oxide, vinyl chloride, propylene oxide, nitromethane, 2-nitropropane, vinyl acetate, ethylbenzene
Room Air Samples (RAS) - Metals | Clinic Visit (JUUL/VUSE: 2 days and 2 overnights; conventional cigarette: 1 day and 1 overnight)
  Absolute change from baseline in metal levels in the room air when subjects use JUUL or VUSE Solo over 4-hour prescribed conditions and JUUL, VUSE Solo, or conventional cigarettes over 4-hour ad libitum conditions. Metals include: arsenic, cadmium, chromium, nickel.
Room Air Samples (RAS) - PM2.5 Particles | Clinic Visit (JUUL/VUSE: 2 days and 2 overnights; conventional cigarette: 1 day and 1 overnight)
  Absolute change from baseline levels of PM2.5 particles in room air when subjects use JUUL or VUSE Solo over 4-hour prescribed conditions and JUUL, VUSE Solo, or conventional cigarettes over 4-hour ad libitum conditions.
Room Air Samples (RAS) - PM10 Particles | Clinic Visit (JUUL/VUSE: 2 days and 2 overnights; conventional cigarette: 1 day and 1 overnight)
  Absolute change from baseline levels of PM10 particles in room air when subjects use JUUL or VUSE Solo over 4-hour prescribed conditions and JUUL, VUSE Solo, or conventional cigarettes over 4-hour ad libitum conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Couroux, MD, Principal Investigator — Inflamax Research
Locations (1):
- Inflamax Research Limited, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bam TS, Bellew W, Berezhnova I, Jackson-Morris A, Jones A, Latif E, Molinari MA, Quan G, Singh RJ, Wisotzky M; Tobacco Control Department International Union Against Tuberculosis and Lung Disease. Position statement on electronic cigarettes or electronic nicotine delivery systems. Int J Tuberc Lung Dis. 2014 Jan;18(1):5-7. doi: 10.5588/ijtld.13.0815. No abstract available. PMID 24365545
- [Background] Schober W, Szendrei K, Matzen W, Osiander-Fuchs H, Heitmann D, Schettgen T, Jorres RA, Fromme H. Use of electronic cigarettes (e-cigarettes) impairs indoor air quality and increases FeNO levels of e-cigarette consumers. Int J Hyg Environ Health. 2014 Jul;217(6):628-37. doi: 10.1016/j.ijheh.2013.11.003. Epub 2013 Dec 6. PMID 24373737
- [Background] Schripp T, Markewitz D, Uhde E, Salthammer T. Does e-cigarette consumption cause passive vaping? Indoor Air. 2013 Feb;23(1):25-31. doi: 10.1111/j.1600-0668.2012.00792.x. Epub 2012 Jul 2. PMID 22672560
- [Background] Czogala J, Goniewicz ML, Fidelus B, Zielinska-Danch W, Travers MJ, Sobczak A. Secondhand exposure to vapors from electronic cigarettes. Nicotine Tob Res. 2014 Jun;16(6):655-62. doi: 10.1093/ntr/ntt203. Epub 2013 Dec 11. PMID 24336346
- [Background] Chang H. Research gaps related to the environmental impacts of electronic cigarettes. Tob Control. 2014 May;23 Suppl 2(Suppl 2):ii54-8. doi: 10.1136/tobaccocontrol-2013-051480. PMID 24732165
- [Background] Liu J, Liang Q, Oldham MJ, Rostami AA, Wagner KA, Gillman IG, Patel P, Savioz R, Sarkar M. Determination of Selected Chemical Levels in Room Air and on Surfaces after the Use of Cartridge- and Tank-Based E-Vapor Products or Conventional Cigarettes. Int J Environ Res Public Health. 2017 Aug 28;14(9):969. doi: 10.3390/ijerph14090969. PMID 28846634
- [Background] Hess IM, Lachireddy K, Capon A. A systematic review of the health risks from passive exposure to electronic cigarette vapour. Public Health Res Pract. 2016 Apr 15;26(2):2621617. doi: 10.17061/phrp2621617. PMID 27734060
- [Background] ANSI/ASHRAE Standard 62.1-2016. Ventilation for Acceptable Indoor Air Quality. American Society of Heating, Refrigerating and Air-Conditioning Engineers, Inc.